CLINICAL TRIAL: NCT01676922
Title: Prospective Non-interventional Study to Collect Data on the Use of Avastin and Conventional Chemotherapy for the Treatment of Previously Untreated Metastatic Colorectal Cancer in Patients >/= 70 Years
Brief Title: An Observational Study of Avastin and Conventional Chemotherapy in Patients >/= 70 Years of Age With Previously Untreated Metastatic Colorectal Cancer (AVAPLUS)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27768
Record Dates: First submitted 2012-08-27; First posted 2012-08-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the use of Avastin (bevacizumab) and conventional chemotherapy in patients >/= 70 years of age with previously untreated metastatic colorectal cancer. Data will be collected from each patient from initiation of treatment until disease progression occurs (minimum follow-up 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/ 70 years of age
* Previously untreated metastatic colorectal cancer
* Patient considered suitable to receive chemotherapy with or without Avastin

Exclusion Criteria:

* Participation in any other clinical trial or study with the exception of participation in registries

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients >/= 70 years of age with previously untreated metastatic colorectal cancer suitable to receive chemotherapy with or without Avastin
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2011-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Treatment duration in patients receiving chemotherapy with Avastin as first-line therapy in daily clinical practice | approximately 24 months

SECONDARY OUTCOMES:
Treatment duration in patients receiving chemotherapy alone as first-line therapy in daily clinical practice | approximately 24 months
Safety: Incidence of adverse events/adverse events of special interest | approximately 24 months
Clinical/demographic patient characteristics at baseline | approximately 24 months
Dosage/regimen | approximately 24 months
Correlation between Comprehensive Geriatric Assessment (CGA) scores and initial treatment | approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- Belgium (31):
  - Aalst
  - Antwerp
  - Assebroek
  - Bonheiden
  - Bornem
  - Brasschaat
  - Bruges
  - Brussels
  - Ghent
  - Haine-Saint-Paul
  - Hasselt
  - Hornu
  - Ieper
  - Kortrijk
  - Leuven
  - Lier
  - Liège
  - Mechelen
  - Mons
  - Mont-godinne
  - Namur
  - Ostend
  - Oudenaarde
  - Roeselare
  - Ronse
  - Seraing
  - Sint-Niklaas
  - Tongeren
  - Turnhout
  - Verviers
  - Wilrijk